CLINICAL TRIAL: NCT04129931
Title: PrecISE (Precision Interventions for Severe and/or Exacerbation-Prone Asthma) Network Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-1681; 5U24HL138998-03 (NIH)
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — clazakizumab; Broncho-Vaxom; Imatinib Mesylate; cavosonstat

STUDY DESIGN:
Intervention Model Description: Treatment sequence will be randomly assigned as either test treatment followed by matching placebo or vice-versa.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Medium Chain Triglycerides (MCT) (Experimental): Participants in this arm will receive Medium Chain Triglycerides (MCT) powder packets (10 g each) at each treatment visit at any point in the study. Participants will mix 1-2 packets of MCT supplement powder into liquids or semi-solid food and ingest 3 times a day during the 16-week treatment period. Participants will be randomized to the treatment sequence and will receive either the active MCT or the matching placebo first or vice versa.
  Interventions: Drug: MCT; Other: Placebo
- Clazakizumab (Experimental): Participants randomized to this arm will receive a 12.5 mg dose of Clazakizumab via a subcutaneous injection at every study visit, every 4 weeks, during the 16-week treatment period at any point in the study. Participants will be randomized to the treatment sequence and will receive either the active Clazakizumab or the matching placebo first or vice versa.
  Interventions: Drug: Clazakizumab; Other: Placebo
- Broncho-Vaxom (Experimental): Participants randomized to this arm will receive 7 mg of Broncho-Vaxom once a day on an empty stomach for the 16-week treatment period duration at any point in the study. Participants will be randomized to the treatment sequence and will receive either the active Broncho-Vaxom or the matching placebo first or vice versa.
  Interventions: Drug: Broncho-Vaxom; Other: Placebo
- Imatinib (Experimental): At any point in the study, participants randomized to this arm will take two 100 mg Imatinib tablets orally once a day with a meal and an 8 oz glass of water for 2 weeks. Participants will then take four 100 mg tablets once a day with a meal and an 8 oz glass of water for 14 weeks. Participants will be randomized to the treatment sequence and will receive either the active Imatinib or the matching placebo first or vice versa.
  Interventions: Drug: Imatinib Mesylate; Other: Placebo
- Cavosonstat (Experimental): Participants randomized to this arm will take one 50 mg Cavosonstat capsule orally twice a day for the 16-week treatment period duration at any point in the study. Participants will be randomized to the treatment sequence and will receive either the active Cavosonstat or the matching placebo first or vice versa.
  Interventions: Drug: Cavosonstat; Other: Placebo

INTERVENTIONS:
Drug: MCT — Mix 1-2 packets, as instructed by a physician, into liquid or food three times daily
  Other Names: Breathe Better Diet (BBD)
  Arms: Medium Chain Triglycerides (MCT)
Drug: Clazakizumab — 12.5 mg subcutaneous injection given once every 4 weeks for 16 weeks. Lab driven dose reductions will be made based on safety lab data. If criteria are met for dose reduction, the participant will be reduced to a 6.25 mg dose.
  Other Names: Anti-interleukin 6 monoclonal antibody; Anti-IL-6 mAb; BMS-945429; ALD518
  Arms: Clazakizumab
Drug: Broncho-Vaxom — 7 mg taken orally once a day, on an empty stomach, for 16 weeks
  Other Names: OM-85 BV VEGETAL
  Arms: Broncho-Vaxom
Drug: Imatinib Mesylate — Two 100 mg tablets orally once a day with a meal and an 8 oz glass of water for 2 weeks. If the drug is well tolerated, participants will titrate up to four 100 mg tablets once a day with a meal and an 8 oz glass of water for 14 weeks. Safety labs will be collected at each study visit to monitor the tolerability of each participant.
  Other Names: Gleevec; Zoleta; Glivec; Ziatir
  Arms: Imatinib
Drug: Cavosonstat — 50 mg capsule orally twice a day for 16 weeks.
  Other Names: N91115
  Arms: Cavosonstat
Other: Placebo — MCT Matching Placebo: MCT matching placebo packets. Mix 1-2 packets, as instructed by a physician, into liquid or food three times daily
  Clazakizumab Matching Placebo: 12.5 mg subcutaneous saline injection given once every 4 weeks for 16 weeks.
  Broncho-Vaxom Matching Placebo: 7 mg matching placebo taken orally once a day on an empty stomach for 16 weeks
  Imatinib Matching Placebo: Two 100 mg placebo tablets orally once a day with a meal and an 8 oz glass of water for 2 weeks. Then four 100 mg placebo tablets once a day with a meal and an 8 oz glass of water for 14 weeks.
  Cavosonstat Matching Placebo: 50 mg matching placebo capsule orally twice a day for 16 weeks.

SUMMARY:
The primary objective of this study is to evaluate several interventions given to participants with severe asthma. Interventions are administered in a crossover manner with 16-week treatment periods followed by 8 to 16 week washout.

DETAILED DESCRIPTION:
PrecISE is a clinical study sponsored by the U.S. National Heart, Lung, and Blood Institute (NHLBI) to investigate several treatments for severe asthma. PrecISE will enroll 600 adults and teenagers (ages 12 years and older) with severe asthma who have symptoms that are not well-controlled on high dose of inhaled corticosteroids including those who have frequent asthma attacks. Each person who agrees to enroll in the PrecISE study will receive several treatments for research purposes based on their type of severe asthma.

The goal of PrecISE is to understand how to treat different types of severe asthma, by using precision medicine. Precision medicine is an approach that targets treatments to defined subgroups of patients who share similar characteristics, for example, patients with a certain genetic variation or patients with high number of blood eosinophils.

Researchers from over 30 locations across the US are involved in PrecISE.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Started willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, age ≥ 12 years
4. No change in asthma medications for the past 2 months and use of medium or high dose inhaled corticosteroids (ICS) (defined by Table 1A) + an additional asthma controller/biologic (defined in Tables 1B and 1C). Participants entered into the run-in on medium dose ICS will be switched to high dose ICS. They must meet all entry criteria at the time of randomization including the criteria for uncontrolled asthma as assessed by symptoms during the two weeks prior to the randomization.
5. Baseline poor or uncontrolled asthma, defined as meeting at least one of the following:

   1. FEV1 <80% predicted (for adults ≥18) or FEV1<90% (pediatric participants <18) AND with 12% bronchodilator reversibility
   2. Poor symptom control - Asthma Control Questionnaire ( ACQ-6) Score ≥1.5
   3. ≥1 exacerbation defined as a documented burst of systemic corticosteroids (>3 days for adults and adolescents or >1 day for adolescents treated with dexamethasone) in prior year for those not receiving chronic OCS or an increase in >50% of baseline corticosteroid dose for ≥3 days in those receiving chronic OCS.

      * For patients on a biologic agent, at least one asthma exacerbation must have occurred at least 2 months after the initiation of the biologic agent. The definition of acceptable documentation for asthma exacerbations can be found in Section 6.5.3.
6. Evidence of asthma demonstrated by either bronchodilator reversibility or methacholine responsiveness either during the run-in or by historical evidence of either criterion if testing was performed under the same standards of the PrecISE Network at a PrecISE recruitment center. These criteria are defined as:

   1. An increase in FEV1 ≥12% (and 200 ml) after up to 8 puffs of albuterol OR
   2. Positive methacholine defined as PC20 ≤16 mg/ml, or PD20 ≤400 mcg/ml
7. Agreement to adhere to Lifestyle Considerations (see Section 5.4) throughout study duration
8. Owns a device compatible with the eDiary system used for CompEx, that is, an iOS 11+ device such as iPhone, iPad or iPod, or a smartphone or tablet running on Android 5.0+

Exclusion Criteria:

1. Current participation in an interventional trial (e.g. drugs, diets, etc.)
2. Enrollment in a clinical trial where the study medication was administered within the past 60 days or within 5 half-lives (whichever is greater)
3. Physician diagnosis of other chronic pulmonary disorders associated with asthma-like symptoms, including, but not limited to, cystic fibrosis (CF), chronic obstructive pulmonary disease (COPD), chronic bronchitis, emphysema, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways
4. Receiving one or more immune-modulating therapies for diseases other than asthma
5. Receiving methotrexate, mycophenolate (CellCept®), or azathioprine (Imuran®)
6. Receiving aero allergen immunotherapy and not on at least 3 months of maintenance allergen immunotherapy
7. Underwent a bronchial thermoplasty within the last two years
8. Born before 35 weeks of gestation
9. Uncontrolled hypertension, defined as systolic blood pressure >160 mm/Hg, or diastolic blood pressure >100 mm/Hg
10. History of malignancy except non-melanoma skin cancer within the last five years
11. History of smoking

    1. If <30 years old: Smoked for ≥5 pack-years*

       * Can still be enrolled if <30, smoked <5 5 pack years and none in past year, and normal (negative) urine cotinine
    2. If 30-39 years old: Smoked for ≥10 pack years

       * Can still be enrolled if ≥30, smoked <10 pack years and none in past year, provided participant demonstrates a normal (negative) urine cotinine
    3. If ≥40 years old: Smoked ≥15 pack years

       * Can still be enrolled if ≥40 years old, smoked <15 pack years and none in the last year, provided participant demonstrates normal (negative) urine cotinine. Patients with a smoking history of ≥10 to <15 pack years will also need to demonstrate a normal Diffusing Capacity for Carbon Monoxide (DLCO) (>70% predicted) * Smoking equivalent pack years. One pack of cigarettes a day for 1 year is equivalent to:

    <!-- -->

    1. 1 cigar or pipe per day for 1 year
    2. Smoked hookah or shisha =1 session per day for 1 year
    3. Vaped e-cigarettes =0.5 mLs e-liquid per day for 1 year, or =1 cartridge/tank/pod per day for 1 year
    4. 1 use of marijuana per day for 1 year
12. Active use of any inhalant >1 time per month in the past year

    1. Active smoking of conventional tobacco, inhaling of marijuana or other drugs, or vaping of e-cigarettes or vape pods >1 time per month in the past year
    2. Any form of tobacco qualifies, such as: 1 cigarette, 1 hookah or shisha sessions, 1 cigar, 1 pipe, etc.
    3. Any electronic (e)-device included: e-cigarette e-cig, mod, vape pen, JUUL vaping device, e-cigar, e-hookah, e-pipe, vape pods, etc.
    4. Any form of inhaled marijuana, including smoking marijuana leaves or inhaling THC (tetrahydrocannabinol) via e-cigarette or device
13. Substance abuse within the last year
14. Unwillingness to practice medically acceptable birth control or complete abstinence during the study, current pregnancy, or lactation. Medically acceptable birth control/abstinence is defined as:

    1. Career, lifestyle, or sexual orientation precludes intercourse with a male partner
    2. For those in a monogamous relationship that precludes sexual activity with other partners, one of the sexual partners has been sterilized by vasectomy (in males) or hysterectomy and/or bilateral salpingo-oophorectomy (in females)
    3. Use of highly effective methods of birth control defined as those, alone or in combination, that result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Contraception should be used for at least 1 month prior to screening, throughout study participation and for an additional 16 weeks after the end of the final test treatment.

       * Pregnancy tests will be given to each female participant prior to study enrollment and at each clinic visit
       * Each male participant will agree to inform his sexual partner(s) of the potential for harm to an unborn child. If a sexual partner becomes pregnant while he is participating in the study, he will notify study staff within 24 hours of receiving medical confirmation. His partner will be advised to promptly notify her doctor
       * Any pregnancy (of a participant or a partner) will be monitored for adverse events with respect to pregnancy outcome until one month after birth.
15. Requirement for daily systemic corticosteroids above 10 mg of prednisone (or equivalent) per day for the past 2 months
16. Respiratory infection within 1 month of screening
17. Intubation for asthma in the last 12 months
18. Use of warfarin, current or last 30 days
19. Any clinically significant abnormal findings in the history, physical examination, vital signs, electrocardiogram, hematology or clinical chemistry during run-in period, which in the opinion of the site investigator, may put the participant at risk because of his/her participation in the study, or may influence the results of the study, or the participant's ability to complete the entire duration of the study
20. Additional exclusions for specific interventions (and not for others) are listed in the Appendices I-VI, Section 5.2

Safety Exclusion Criteria:

Participants who meet the following criteria will be excluded from the study:

1. Hemoglobin <10 g/dL
2. Absolute Neutrophil Count (ANC) <1000/µl for black participants, <1500/µl for other participants
3. Lymphocytes <500/µl
4. Platelet count <100,000/µl
5. Alanine Transaminase (ALT)/Aspartate Aminotransferase (AST) >2x upper limits of normal (ULN)
6. Bilirubin ≥2x ULN
7. Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 sq m
8. Positive Human Immunodeficiency Virus, Types 1 & 2 (HIV 1&2) Ab/Ag immunoassay followed by a confirmatory positive test (Geenius™ HIV-1/HIV-2 antibody differentiation immunoassay)
9. Positive Hepatitis B surface Ag (active infection) or Hepatitis B core total antibody (marker of past infection that could reactivate)
10. Positive Hepatitis C RNA test following positive Hepatitis C Antibody
11. EKG with significant clinical findings

A positive QuantiFERON-TB (tuberculosis) Gold test requires further screening. A participant may be included in PrecISE if at least one of the following criteria are met:

1. A chest radiograph (CXR) done within the last six months of the test that shows no evidence of active TB
2. A chest CT scan done within the last six months of the test that shows no evidence of active TB
3. Documentation of adequate treatment for latent TB In cases of an indeterminate QuantiFERON-TB test result, a second blood specimen must be drawn. A chest x-ray is not required if the participant has a negative QuantiFERON-TB Gold test.

Comorbid Conditions:

Comorbidities are commonly present in severe asthma. Specific questionnaires will be used to identify common comorbidities as follows:

1. Sleep apnea: STOP-BANG
2. GERD (GERD- Questionnaire)
3. VCD (Pittsburgh vocal cord dysfunction index)
4. Chronic Rhinitis Sinusitis (Sinonasal questionnaire-SNQ5)
5. Depression-Anxiety (Hospital anxiety and depression Scale: HADS) These questionnaires are best used as screening tools. As such they typically have high sensitivity but relatively low specificity. Many of their symptoms overlap with the symptoms reported by participants with asthma who do not suffer from these conditions. Therefore, participants who meet the established cut offs for these questionnaires will need to be evaluated by the investigator to consider the clinical significance of the positive questionnaire based on history and physical and available testing. The investigator will need to judge the presence, severity and control of a specific condition and determine if it is sufficiently controlled to keep the participant in the PrecISE protocol. If the comorbid condition(s) is/are not adequately controlled, the investigator may refer the participant for further evaluation/treatment, prior to enrollment in PrecISE. Rescreening is permitted (after at least four weeks) to determine if the participant is able to move forward in PrecISE once the comorbid condition(s) is/are under adequate control. It is expected that some of the participants may also have other conditions such as cardiovascular disease, diabetes and obesity. These should be evaluated clinically as part of the complete history and physical done at initial evaluation. Their inclusions should be based on the investigator clinical judgement in line with good clinical practice principles.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1) percent predicted | Measured at 16 weeks after the start of treatment.
  Assessed prior to bronchodilator administration. Efficacy analyses will compare the end-of-period outcome values between test treatment and placebo.
The Juniper Asthma Control Questionnaire (ACQ-6) | Measured at 16 weeks after the start of treatment.
  Asthma symptom control is assessed via ACQ-6, the average score of these six items (range 0-6). The seven-point response scale: 0 = 'totally controlled' and 6 = 'severely uncontrolled'. Negative change from baseline values indicate improved asthma control. Efficacy analyses will compare the end-of-period outcome values between test treatment and placebo.
CompEx events | Assessed over 16 weeks of treatment
  CompEx is a composite outcome specific to asthma that combines clinically-relevant deteriorations captured by diary events with exacerbations. CompEx events include exacerbations and deterioration events defined based on daily recordings of peak expiratory flow (PEF) morning/evening (L/min), reliever use morning/evening (doses), symptoms morning/evening (score 0-3) from twice-daily recordings. Participants will be asked to describe their morning and symptoms using the following scale: 0-No symptoms to report, 3-I could not sleep because of my asthma/I could not perform my normal activities because of my asthma.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) pre-bronchodilation | Measured at 16 weeks after the start of treatment.
  Assessed prior to bronchodilator administration
FEV1 post-bronchodilation | Measured at 16 weeks after the start of treatment.
  Assessed after bronchodilator administration.
Time to first exacerbation | Assessed over 16 weeks of treatment
Symptom free days | Assessed over 16 weeks of treatment
Asthma free days | Assessed over 16 weeks of treatment
Healthcare utilization | Assessed over 16 weeks of treatment
  Asthma-specific Emergency Department visits, asthma-specific hospital admissions, and asthma-specific ICU admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Ivanova, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (29):
- United States (29):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of Arizona Tucson, Tucson, Arizona
  - University of California Davis, Sacramento, California
  - University of California San Diego: Airway Research & Clinical Trials Center, San Diego, California
  - University of California San Diego: La Jolla Altman Clinical Translation Research Institute, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Northwestern Universtiy, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Israel E, Reddel HK. Severe and Difficult-to-Treat Asthma in Adults. N Engl J Med. 2017 Sep 7;377(10):965-976. doi: 10.1056/NEJMra1608969. No abstract available. PMID 28877019
- [Background] Woodcock J, LaVange LM. Master Protocols to Study Multiple Therapies, Multiple Diseases, or Both. N Engl J Med. 2017 Jul 6;377(1):62-70. doi: 10.1056/NEJMra1510062. No abstract available. PMID 28679092
- [Background] Fuhlbrigge AL, Bengtsson T, Peterson S, Jauhiainen A, Eriksson G, Da Silva CA, Johnson A, Sethi T, Locantore N, Tal-Singer R, Fageras M. A novel endpoint for exacerbations in asthma to accelerate clinical development: a post-hoc analysis of randomised controlled trials. Lancet Respir Med. 2017 Jul;5(7):577-590. doi: 10.1016/S2213-2600(17)30218-7. Epub 2017 Jun 2. PMID 28583396
- [Background] Phipatanakul W, Mauger DT, Sorkness RL, Gaffin JM, Holguin F, Woodruff PG, Ly NP, Bacharier LB, Bhakta NR, Moore WC, Bleecker ER, Hastie AT, Meyers DA, Castro M, Fahy JV, Fitzpatrick AM, Gaston BM, Jarjour NN, Levy BD, Peters SP, Teague WG, Fajt M, Wenzel SE, Erzurum SC, Israel E; Severe Asthma Research Program. Effects of Age and Disease Severity on Systemic Corticosteroid Responses in Asthma. Am J Respir Crit Care Med. 2017 Jun 1;195(11):1439-1448. doi: 10.1164/rccm.201607-1453OC. PMID 27967215
- [Background] Waljee AK, Rogers MA, Lin P, Singal AG, Stein JD, Marks RM, Ayanian JZ, Nallamothu BK. Short term use of oral corticosteroids and related harms among adults in the United States: population based cohort study. BMJ. 2017 Apr 12;357:j1415. doi: 10.1136/bmj.j1415. PMID 28404617
- [Background] Moore WC, Meyers DA, Wenzel SE, Teague WG, Li H, Li X, D'Agostino R Jr, Castro M, Curran-Everett D, Fitzpatrick AM, Gaston B, Jarjour NN, Sorkness R, Calhoun WJ, Chung KF, Comhair SA, Dweik RA, Israel E, Peters SP, Busse WW, Erzurum SC, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Identification of asthma phenotypes using cluster analysis in the Severe Asthma Research Program. Am J Respir Crit Care Med. 2010 Feb 15;181(4):315-23. doi: 10.1164/rccm.200906-0896OC. Epub 2009 Nov 5. PMID 19892860
- [Background] Peters SP, Kunselman SJ, Icitovic N, Moore WC, Pascual R, Ameredes BT, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Craig T, Denlinger L, Engle LL, DiMango EA, Fahy JV, Israel E, Jarjour N, Kazani SD, Kraft M, Lazarus SC, Lemanske RF Jr, Lugogo N, Martin RJ, Meyers DA, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Chinchilli VM, Bleecker ER; National Heart, Lung, and Blood Institute Asthma Clinical Research Network. Tiotropium bromide step-up therapy for adults with uncontrolled asthma. N Engl J Med. 2010 Oct 28;363(18):1715-26. doi: 10.1056/NEJMoa1008770. Epub 2010 Sep 19. PMID 20979471
- [Background] Lemanske RF Jr, Mauger DT, Sorkness CA, Jackson DJ, Boehmer SJ, Martinez FD, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Covar RA, Guilbert TW, Larsen G, Morgan WJ, Moss MH, Spahn JD, Taussig LM; Childhood Asthma Research and Education (CARE) Network of the National Heart, Lung, and Blood Institute. Step-up therapy for children with uncontrolled asthma receiving inhaled corticosteroids. N Engl J Med. 2010 Mar 18;362(11):975-85. doi: 10.1056/NEJMoa1001278. Epub 2010 Mar 2. PMID 20197425
- [Background] Sorkness CA, Lemanske RF Jr, Mauger DT, Boehmer SJ, Chinchilli VM, Martinez FD, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Bloomberg GR, Covar RA, Guilbert TW, Heldt G, Larsen G, Mellon MH, Morgan WJ, Moss MH, Spahn JD, Taussig LM; Childhood Asthma Research and Education Network of the National Heart, Lung, and Blood Institute. Long-term comparison of 3 controller regimens for mild-moderate persistent childhood asthma: the Pediatric Asthma Controller Trial. J Allergy Clin Immunol. 2007 Jan;119(1):64-72. doi: 10.1016/j.jaci.2006.09.042. Epub 2006 Nov 30. PMID 17140647
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Fitzpatrick AM, Szefler SJ, Mauger DT, Phillips BR, Denlinger LC, Moore WC, Sorkness RL, Wenzel SE, Gergen PJ, Bleecker ER, Castro M, Erzurum SC, Fahy JV, Gaston BM, Israel E, Levy BD, Meyers DA, Teague WG, Bacharier LB, Ly NP, Phipatanakul W, Ross KR, Zein J, Jarjour NN. Development and initial validation of the Asthma Severity Scoring System (ASSESS). J Allergy Clin Immunol. 2020 Jan;145(1):127-139. doi: 10.1016/j.jaci.2019.09.018. Epub 2019 Oct 8. PMID 31604088
- [Background] de Wit HM, Te Groen M, Rovers MM, Tack CJ. The placebo response of injectable GLP-1 receptor agonists vs. oral DPP-4 inhibitors and SGLT-2 inhibitors: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Jul;82(1):301-14. doi: 10.1111/bcp.12925. Epub 2016 Apr 22. PMID 26935973
- [Background] Dutile S, Kaptchuk TJ, Wechsler ME. The placebo effect in asthma. Curr Allergy Asthma Rep. 2014 Aug;14(8):456. doi: 10.1007/s11882-014-0456-2. PMID 24951239
- [Background] Wise RA, Bartlett SJ, Brown ED, Castro M, Cohen R, Holbrook JT, Irvin CG, Rand CS, Sockrider MM, Sugar EA; American Lung Association Asthma Clinical Research Centers. Randomized trial of the effect of drug presentation on asthma outcomes: the American Lung Association Asthma Clinical Research Centers. J Allergy Clin Immunol. 2009 Sep;124(3):436-44, 444e1-8. doi: 10.1016/j.jaci.2009.05.041. Epub 2009 Jul 25. PMID 19632710
- [Background] Zhu R, Zeng D, Kosorok MR. Reinforcement Learning Trees. J Am Stat Assoc. 2015;110(512):1770-1784. doi: 10.1080/01621459.2015.1036994. Epub 2015 Apr 16. PMID 26903687
- [Background] Zhao Y, Zeng D, Rush AJ, Kosorok MR. Estimating Individualized Treatment Rules Using Outcome Weighted Learning. J Am Stat Assoc. 2012 Sep 1;107(449):1106-1118. doi: 10.1080/01621459.2012.695674. PMID 23630406
- [Background] Murphy SA. An experimental design for the development of adaptive treatment strategies. Stat Med. 2005 May 30;24(10):1455-81. doi: 10.1002/sim.2022. PMID 15586395
- [Background] Gallo P., DeMets D., LaVange L. (2014) Considerations for Interim Analyses in Adaptive Trials, and Perspectives on the Use of DMCs. In: He W., Pinheiro J., Kuznetsova O. (eds) Practical Considerations for Adaptive Trial Design and Implementation. Statistics for Biology and Health. Springer, New York, NY
- See also: US Food and Drug Administration. Draft Guidance for Industry: Adaptive Designs for Clinical Trials of Drugs and Biologics. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/adaptive-design-clinical-trials-drugs-and-biologics
- See also: US Food and Drug Administration. Guidance for Clinical Trial Sponsors on Establishment and Operation of Clinical Trial Data Monitoring Committees — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/establishment-and-operation-clinical-trial-data-monitoring-committees
- See also: ICH (International Conference on Harmonization) Harmonized Guideline E9 Statistical Principles for Clinical Trials — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/e9-statistical-principles-clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-10-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04129931/ICF_000.pdf